CLINICAL TRIAL: NCT03122626
Title: Increasing Access to Community-based Task-oriented Exercise Programs Through Healthcare-recreation Partnerships to Improve Function Post-stroke: Feasibility of a 2-group Randomized Controlled Trial Protocol
Brief Title: Does a Group, Task-oriented Community-based Exercise Program Improve Everyday Function in People With Stroke?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other); Heart and Stroke Foundation of Canada (Other); University of Western Ontario, Canada (Other); Ontario Stroke Network (Other); Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Principal Investigator, Dr. Nancy Salbach, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G-16-00013979
Record Dates: First submitted 2017-04-10; First posted 2017-04-21 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Stroke; Balance; Mobility Limitation; Activities of Daily Living
Keywords: stroke; community-based exercise program; task-oriented exercise; group exercise program; healthcare-recreation partnership; randomized controlled pilot trial; mixed methods
MeSH Terms: conditions — Stroke; Mobility Limitation | interventions — Movement; Exercise; Time

STUDY DESIGN:
Intervention Model Description: A 2-group randomized controlled trial in which participants are assigned to immediate or delayed participation in a community exercise program
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be unaware of group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The intervention is a group, task-oriented exercise program involving two 1-hour exercise classes per week for 12 weeks. The class involves a seated warm-up, repetitive, progressive practice of functional balance and mobility tasks, and a seated cool down. The warm-up consists of active range-of-motion exercises, aerobic exercise, leg loading, stretching, and sit-to-stand training. The cool-down involves exercises with an emphasis on stretching and relaxation. Tasks are organized in a 3-station circuit completed by participants grouped by overall ability: Superstation 1: walking, aerobic training, and wall work (standing and reaching, wall push-ups); Superstation 2: standing weight shifts, coordinated with stepping and lunging; and Superstation 3: tap-ups, step-ups, and heel/toe raises, hamstring curls, marching-on-the-spot, and mini-squats. Participants are instructed to be physically active by walking in their neighbourhood, practicing the program exercises, or using the stairs.
  Interventions: Behavioral: Together in Movement and Exercise (TIME) Program
- Wait-listed Control Group (No Intervention): The control group will receive usual care which will be monitored and is expected to consist of provision of a home exercise program and information on community resources according to current best practices. At the end of the study period, participants in the control group will be offered to participate in the 3-month exercise program.

INTERVENTIONS:
Behavioral: Together in Movement and Exercise (TIME) Program — The TIME program is an evidence-based, standardized, progressive, licensed exercise program developed by physical therapists at the Toronto Rehabilitation Institute-University Health Network.
  Arms: Experimental Group

SUMMARY:
After a stroke, people find it difficult to perform everyday activities independently, like getting dressed, preparing meals, and shopping, limiting their independence and requiring the assistance of a family member, friend or a home care worker. Losing one's independence can decrease quality of life. Functional exercise classes run by physical therapists where people with stroke practice getting in and out of a chair, stepping, and walking, can improve the ability to balance, walk, and do everyday activities. These classes are not commonly available in community centres, mainly because fitness instructors do not receive training in how to run exercise classes for people with stroke. Therefore there is a need to make these functional exercise programs available in local community centres.

The objective of this project is to test procedures for running a large study to see whether people with stroke improve their ability to do everyday activities after participating in functional group exercise classes for 12 weeks in local community centres. If ability to do everyday activities improves, the investigators wish to see if the improvement is still present 3, 6 and 9 months later. Physical therapists at a nearby hospital will teach fitness instructors how to run the exercise class, help out during the classes, and answer questions by email or phone. Before conducting the larger Canada-wide study, it is important to determine the interest in such a program, the acceptability of the evaluations and the costs associated with the program, the degree of improvements resulting from the program, and if fitness instructors are able to run the program as planned.

In Toronto, London and Pembroke, Canada, managers at a hospital and a nearby recreation centre have agreed to help run the exercise program. A recruiter will ask people with stroke who can walk and are being discharged home from the hospital whether they can be called about the study. People with stroke and a caregiver who agree to participate in the study will complete four evaluations when they enter the study, and 3, 6, and 12 months later. At each evaluation, people with stroke will perform tests of balance and walking, and complete questionnaires about their mood, participation in valued activities, and quality of life. After the first evaluation, the investigators will use a process like flipping a coin, to see if the person with stroke will begin the exercise program immediately or 12 months later. The investigators will call people each month to ask if a fall occurred. The investigators will interview exercise participants, family members and hospital/recreation staff at the end of the study to ask about the experiences.

This project is unique because the program combines the expert knowledge and skills of physical therapists and fitness instructors. The exercise program involves practicing everyday movements, making the exercises easy for fitness instructors and people with stroke to learn. Each exercise has multiple levels of difficulty so the instructor can adapt exercises to how the person is feeling. The exercise program does not require expensive equipment (e.g. chairs, stepping stools) and therefore can be offered in most community centres. Finally, an extensive network of hospitals providing stroke care and community centres run by recreation organizations exists in Canada. Thus, if this program is beneficial, it could easily be made widely available.

With the number of Canadians living with the consequences of stroke increasing every year, access to a functional exercise programs in local community centres will improve their ability to function and live independently in the community and reduce the burden on family or caregivers and on the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke recorded in the health record;
* Age ≥ 18 years;
* Living at home for at least 3 months;
* Ability to walk a minimum of 10 metres with or without walking aids without assistance from another person;
* Ability to follow verbal instructions or demonstrations of the exercises;
* Ability to speak and read English; and
* Willingness to obtain medical clearance from a healthcare provider and sign a liability waiver.

Exclusion Criteria:

* Self-reported involvement in another formal exercise or rehabilitation program;
* Conditions or symptoms preventing participation in exercise (e.g., unstable cardiovascular disease, significant joint pain);
* Cognitive or behavioural deficits that would prevent cooperation within a group;
* Self-reported ability to walk more than 20 minutes without a seated rest; and
* Self-reported ability to manage environmental barriers (curbs, ramps, and stairs) with relative ease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Subjective Index of Physical and Social Outcome (SIPSO) | Change from baseline to 3 months.
  10-item, self-report questionnaire. 2 subscales: physical function (5 items), social function (5 items)
Nottingham Extended Activities of Daily Living (NEADL) | Change from baseline to 3 months.
  22-item, self-report performance of instrumental ADL in 4 categories: mobility, kitchen, domestic, and leisure.

SECONDARY OUTCOMES:
Barthel Index | 5 Baseline, 3 months, 6 months, and 12 months
  10-item, self-report or objective measure to assess level of independence in ability to perform basic activities of daily living
EuroQol five dimensions questionnaire | Baseline, 3 months, 6 months, and 12 months
  5-item, self report questionnaire to assess health utility
Stroke Impact Scale | Baseline, 3 months, 6 months, and 12 months
  59-item, self-report, 8 scales: strength, hand function, activities of daily living, mobility, communication, emotion, memory and thinking, participation.
Berg Balance Test | Baseline, 3 months, 6 months, and 12 months
  14-items, objective measure designed to assess static balance and fall risk in adult populations
Activities-specific Balance Confidence (ABC) Scale | Baseline, 3 months, 6 months, and 12 months
  16-item, self-report; level of confidence in doing activities without losing balance or becoming unsteady
30-second Timed Sit-to-stand Test | Baseline, 3 months, 6 months, and 12 months
  Number of full sit-to-stands as possible in 30 seconds starting from a sitting position in a chair of standard height (43.2 cm) with no arm-rests
6-Minute Walk Test | Baseline, 3 months, 6 months, and 12 months
  Maximum distance walked in 6 minutes (standard encouragement each minute) on a straight 30-metre path.
10-metre Walk Test | Baseline, 3 months, 6 months, and 12 months
  Time taken to walk the middle 10 m of a 14-m walkway at a comfortable and maximum pace
Life Space Assessment questionnaire | Baseline, 3 months, 6 months, and 12 months
  6-item, self-report. Indicate zones of the home, the neighborhood and the community that have been accessed in the past 3 days; the frequency of visit to these places and the use of auxiliary devices/ assistance
Canadian Study of Health and Aging-Clinical Frailty Scale | Baseline, 3 months, 6 months, and 12 months
  Indicates level of frailty of an individual based on impairments in mobility, function and self-rated health
Trail Making Test | Baseline, 3 months, 6 months, and 12 months
  Trails A consists of paper with circled numbers (from 1-25). Participants connect circles in numerical order as fast as possible.
  Trails B consists of paper with circled numbers and letters. Participants connect numbers and letters in order, alternating between numbers and letters.
Geriatric Depression Scale-Short Version | Baseline, 3 months, 6 months, and 12 months
  15-item, self-report. Response options are yes or no. Depressive responses are assigned a score of 1 point. Item-level scores are summed to yield a total score that is used to classify the level of depressive symptoms.
Occurrence of injurious falls | Monthly, Months 1-12
  Participants are provided monthly falls calendar, coordinator contacts monthly to obtain details of any falls
Number of healthcare services utilized | 12 months
  Primary care, Outpatient care, Inpatient care, Community care; Data are routinely collected and can be obtained from the Institute of Clinical and Evaluative Sciences (ICES) 6 months following the study end date
Type of healthcare services utilized | 12 months
  Primary care, Outpatient care, Inpatient care, Community care; Data are routinely collected and can be obtained from the Institute of Clinical and Evaluative Sciences (ICES) 6 months following the study end date
Number of homecare services | Monthly, Months 1-12
  Monthly details of services used
Type of homecare services | Monthly, Months 1-12
  Monthly details of services used
Blood Pressure | Baseline, 3 months, 6 months, and 12 months
  Systolic/Diastolic Pressure
Heart Rate | 0.5 minutes
  Heart rate
Mobility aid type | Baseline, 3 months, 6 months, and 12 months
  Types of mobility aids used
Mobility aid number | Baseline, 3 months, 6 months, and 12 months
  Number of mobility aids used
Stroke characteristic | Baseline
  Date, side and type of stroke
Stroke characteristic date | Baseline
  Date of stroke
Stroke side | Baseline
  Side of brain in which stroke occured
Stroke type | Baseline
  The type of stroke
Sociodemographic data-age | Baseline
  Age in years
Sociodemographic data-sex | Baseline
  Sex
Height | Baseline, 3 months, 6 months, and 12 months
  Height in meters
Weight | Baseline, 3 months, 6 months, and 12 months
  Weight in Kg
Sociodemographic data-employment | Baseline
  Employment Status
Education level | Baseline
  Years of education
Personal income | Baseline
  Category of personal income
Charlson Comorbidity Index | Baseline
  16-item scale to predict mortality. 8 items are given 1 point each, 8 other receive a score depending on the severity of condition
Co-intervention type | Monthly (1-12 months)
  Type of co-intervention
Co-intervention frequency | Monthly (1-12 months)
  Frequency of co-intervention
Caregiver Assistance Scale | Baseline, 3 months, 6 months, and 12 months
  17-item, caregiver self-report Indicates assistance provided to the care recipient in basic and instrumental ADLs and treatment-related activities
Rand | Baseline, 3 months, 6 months, and 12 months
  Emotional well-being and Energy/Fatigue Score, 9-item, self-report; Caregiver's perceived emotional status and energy levels over the past 4 weeks.
Time per week spent caregiving | Baseline, 3 months, 6 months, and 12 months
  Time in hours
Costs report | Bi-weekly (1-3 months)
  Self-reported costs for implementing one 12-week exercise program will be estimated for; healthcare system: salary of physical therapist train and provide consultation to fitness instructors; recreation provider: salary of fitness instructors and program coordinators, marketing, room booking, overhead, and equipment; and program participant: registration fee, transportation, personal health aides, unpaid caregiver's lost salary
Intervention fidelity-activity checklist | Bi-weekly (1-3 months)
  TIME Program activities at Recreation Site-Completed by Fitness Instructors
Intervention feasibility-attendance sheet | Bi-weekly (1-3 months)
  TIME Program attendance at Recreation Site-Completed by Fitness Instructors
PT Evaluation form | Weekly (1-3 months)
  Evaluation conducted by Physical Therapist healthcare partner regarding the adherence to protocol
Adverse events | Weekly (1-3 months)
  Adverse events occurring during the TIME exercise program; completed by fitness instructors

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Salbach, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Department of Physical Therapy, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aravind G, Bashir K, Cameron JI, Bayley MT, Teasell RW, Howe JA, Tee A, Jaglal SB, Hunter S, Salbach NM. What matters to program partners when implementing a community-based exercise program for people post-stroke? A theory-based qualitative study and cost analysis. Front Rehabil Sci. 2023 Aug 14;4:1064206. doi: 10.3389/fresc.2023.1064206. eCollection 2023. PMID 37645234
- [Derived] Aravind G, Bashir K, Cameron JI, Howe JA, Jaglal SB, Bayley MT, Teasell RW, Moineddin R, Zee J, Wodchis WP, Tee A, Hunter S, Salbach NM. Community-based exercise programs incorporating healthcare-community partnerships to improve function post-stroke: feasibility of a 2-group randomized controlled trial. Pilot Feasibility Stud. 2022 Apr 22;8(1):88. doi: 10.1186/s40814-022-01037-9. PMID 35459194